CLINICAL TRIAL: NCT06875856
Title: Comparative Effects of Cailliet and Kendall Exercises on Pain, Functional Movement and Disability in Nonspecific Neck Pain: Randomized Control Trial
Brief Title: Effects of Cailliet and Kendall Exercises in Nonspecific Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0151
Record Dates: First submitted 2025-03-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Nonspecific Neck Pain
Keywords: Cailliet exercises, Kendall exercises, Neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Kendall exercises program (Experimental): Group A will receive Kendall exercises program with baseline treatment.
  Interventions: Other: Kendall exercises
- Group B: Cailliet exercises program (Active Comparator): Group B will receive Cailliet exercises program with baseline treatment.
  Interventions: Other: Cailliet exercises

INTERVENTIONS:
Other: Kendall exercises — 1. Positioning supine with the chin tucked in and lifting the head for 2 to 8 sec to strengthen deep cervical flexors.
  2. Maintaining a sitting posture, with hands on the occipital region, and flexed spine while moving head downwards to stretch cervical extensors, maintaining an upright posture.
  3. Keep the resistance band circling with strong support and stretching it with the upper limbs of both sides so that there is full retraction of the scapula to strengthen retractors of the shoulder.
  4. Stretching the pectoralis major and minor while keeping the patient's hands-on the occipital region and standing behind the patient and pulling both elbows backward to target the bilateral pectoralis muscles
  Arms: Group A: Kendall exercises program
Other: Cailliet exercises — The intervention of group B will include baseline treatment, followed by maneuvers, including: Neck Cailliet exercise using isometric contractions against the prisoner to the maximum that ends with relaxation and continued with stretching. Each posture was maintained for 30 s and 3 sets of 10 repetitions were performed with 3 sessions per week on alternate days for 4 weeks.
  Arms: Group B: Cailliet exercises program

SUMMARY:
Objective of study will be to compare effects of Cailliet and Kendall exercises on pain, functional movement and disability in non-specific neck pain.This randomized clinical trial will be conducted at Good Hands Physiotherapy Clinic, Shahdara Lahore. Sample size of study will be 36. Participants will be randomly divided into two groups Group A and Group B. We will include patients with age group between 25 to 40 years, both genders having localized pain or stiffness in cervical spine for more than 3 months after exclusion of upper limb radiculopathy. Group A will receive Kendall exercises regime and Group B will receive Cailliet exercises regime. Both groups will receive baseline treatment including hot pack and Transcutaneous Electric Nerve Stimulation (TENS). Short term effects would be assessed after treatment for 3 sessions per week on alternate days for 4 weeks. Patients will be assessed by Numeric pain rating scale (NPRS) for pain, Selective Functional Movement Assessment (SFMA) for functional movement and Neck Disability Index (NDI) Urdu version for Disability. Analysis will be done by statistical package for social sciences SPSS 25.

DETAILED DESCRIPTION:
Pain felt in an area circumscribed superiorly by the superior nuchal line, laterally by the neck's lateral borders, and inferiorly by an imagined transverse line passing through the T1 spinous process is defined as neck pain. An acute or chronic cervical and shoulder girdle issue originating from the occiput of the head to the spine of the scapula, with or without limiting cervical range of motion, and unrelated to any past history of infection or fracture can be characterized as non-specific neck pain. One of the most common musculoskeletal issues that impairs general population function and results in disability is neck pain. The cervical spine is a complicated biomechanical system made up of at least 20 pairs of muscles, many of which have similar roles, and countless degrees of flexibility for each joint. However, the etiology and basic pathology of neck pain are still unknown. Around the world, 330 million people experience some form of neck pain with mean estimates of 7.6% prevalence (range, 5.9-38.7%), 37% annual prevalence (range, 16.7-75%), and 48.5% lifetime prevalence (range, 14.2-71%).

There have been contradictory findings from earlier studies about the optimal management of neck pain. While some contend that exercise leads to greater results, others support the efficacy of conventional therapy. Comparing the short-term benefits of the exercise programs designed by Cailliet and Kendall, in order to ascertain which method produces better results in terms of symptom relief and pain reduction. By getting empirical data on the short-term impacts of exercise treatments, the study will advance evidence-based practice. Healthcare practitioners can rely on this information to make well-informed decisions and recommendations because it will provide scientific proof on their safety and efficacy. This will support the use of a more standardized and empirically supported approach in the treatment of generalized neck pain symptoms associated with the neck musculature.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 to 40 years
* Both gender male and female
* Individuals having localized pain or stiffness in spine or both combined between C3 and C7 without upper limb radiculopathy
* Negative Spurling's test, traction test, upper limb tension test, and shoulder abduction test.
* Pain reported on NPRS Moderate score in neck region for more than 3 months
* Neck Disability Index (NDI) score of 0-10 points out of 50 score

Exclusion Criteria:

* Tuberculosis, carcinoma, heart disease, and osteoporosis
* Neural disorders due to prolapsed intervertebral disc
* Any trauma, localized infection or history of surgery in cervical spine region in last 6 months
* Upper motor neuron disease, cervical stenosis, and metabolic diseases in bone and joint
* Hyper flexibility, Open sores
* Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants
* Psychiatric diseases such as phobia/obsession and depression
* Allergy to hot pack

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 weeks
  Pain intensity will be assessed by NPRS. The NPRS has shown to have moderate to high test-retest reliability, ranging from 0.67 to 0.96. The NPRS is shown to have convergent validity between 0.79 and 0.95. The 11-point NPRS (intervals from 0-10) is used to quantify pain intensity; 0 represents no pain, and 10 represent the worst possible agony. Zero indicates absence of pain while 5 indicate moderate pain and 10 indicate unbearable pain. The patient is asked to mark a number on the scale. At the baseline assessment, after 3 weeks and finally at the end of the intervention program, the NPRS scores will be recorded.
Selective Functional Movement Assessment (SFMA) | 4 weeks
  The Selective Functional Movement Assessment (SFMA) is a popular assessment tool used to observe and detect components of dysfunctional movement patterns. The goal of the assessment is to identify impairments throughout the kinetic chain that may be contributing to movement dysfunction and/or pain. Kappa coefficients for intra-rater reliability ranged from 0.21-1.00, while % absolute agreement ranged from 0.64-1.00.
Neck Disability Index (NDI) for disability | 4 weeks
  The neck disability index (NDI) is one of the most commonly used questionnaires to measure neck pain and disability. One study reported that the NDI is a multidimensional construct that measures a broader concept than disability. Each item is scored out of 5 for a maximum total score of 50. Care should be taken in reporting the score as either out of 50 or as a percentage out of 100. A score of 22% or more is considered a significant activities of daily living disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Good hands physiotherapy clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bogduk N. The anatomy and pathophysiology of neck pain. Phys Med Rehabil Clin N Am. 2003 Aug;14(3):455-72, v. doi: 10.1016/s1047-9651(03)00041-x. PMID 12948338